CLINICAL TRIAL: NCT04036344
Title: Buddy Relationships in DermatoloGic Excisions for Skin Cancer ("BRIDGES"): A Trial of One-to-one Peer Support in Patients With Facial Skin Cancers Treated With Mohs Surgery
Brief Title: Buddy Relationships in DermatoloGic Excisions for Skin Cancer
Acronym: BRIDGES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 831704
Record Dates: First submitted 2019-07-25; First posted 2019-07-29 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Skin Cancer Face; Quality of Life; Surgical Wound; Peer Mentorship
MeSH Terms: conditions — Surgical Wound

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Control participants receive treatment for a facial skin cancer with Mohs micrographic surgery (MMS), however, do not receive a peer mentor. Participants complete 3 online Skin Cancer Index (SCI) surveys at enrollment, 1 week follow-up, and 3 month follow-up.
- Mentee - Preoperative Consult (Experimental): Mentees are enrolled at preoperative consultation visit and paired with a peer mentor throughout their treatment of a facial cancer with MMS. Participants have regular contact with their mentor and complete 3 online SCI surveys at enrollment, 1 week follow-up, and 3 month follow-up.
  Interventions: Behavioral: Peer Mentorship Program
- Mentee - Same Day Surgery (Experimental): Mentees are enrolled at same day surgery visit and paired with a peer mentor throughout their treatment of a facial cancer with MMS. Participants have regular contact with their mentor and complete 3 online SCI surveys at enrollment, 1 week follow-up, and 3 month follow-up.
  Interventions: Behavioral: Peer Mentorship Program

INTERVENTIONS:
Behavioral: Peer Mentorship Program — Mentee participants are paired with a previous MMS patient (Mentor) who is greater than 1 year status post MMS treatment for a facial skin cancer. Mentors and mentees maintain regular contact by telephone, video chat, or in-person meetings throughout the mentee's facial skin cancer treatment with MMS.
  Arms: Mentee - Preoperative Consult; Mentee - Same Day Surgery

SUMMARY:
More than 5 million skin cancer surgeries are performed each year in the United States with 80% of tumors appearing on the head and neck. Facial skin cancer diagnosis negatively affects patient quality of life (QOL) and treatment of skin cancer creates visible scars early in the postoperative period, increases anxiety, and impairs social interactions. We believe that these negative psychosocial changes represent an unmet need for additional social support and practical guidance. A one-to-one peer support program designed for skin cancer patients could provide a focused, cost-effective, patient-centered intervention to improve quality of life and increase satisfaction. Comparable one-to-one peer support programs have demonstrated high rates of patient satisfaction and positive QOL outcomes in a wide range of conditions. This prospective peer support program would be the first of its kind for melanoma and keratinocytic skin cancers. Our pilot program was designed in consultation with leading peer mentorship program researchers and we will implement a structured system to match volunteer mentors with patients. Through qualitative and quantitative data, we will evaluate the program's effect on patient QOL at 3 separate intervals: at initial consultation, 1-2 weeks post-surgery, and 3 months post-surgery. We hope that this study will enable us to design and execute a larger multi-center clinical trial in order to establish a best practice for surgeons to usher patients through the postoperative healing process after skin cancer surgery.

DETAILED DESCRIPTION:
Skin cancer is a common, often chronic condition that negatively impacts patient quality of life. Currently, more than 5 million skin cancer surgeries are performed in the United States each year, at a cost of over $8 billion per year. Eighty percent of these tumors occur on the head and neck, anatomic sites most visible to society. Recent studies have demonstrated that patients have reduced concern about the severity and prognosis of their skin cancer in the period immediately following Mohs micrographic surgery (MMS). However, patient QOL related to appearance and social interactions is impaired in the weeks following MMS due to elevated distress regarding post-surgical physical appearance.

One-to-one peer support programs benefit both the patient and the mentor. In one-to-one peer support programs, individuals previously affected by a disease or condition volunteer to provide support to current patients in a loosely structured, mentorship setting. Peer mentors provide mentees with social and emotional support as well as practical guidance on health system navigation. Similar peer mentorship programs with burn patients who had significant changes to outward physical appearance resulted in positive experiences for both mentee and mentor. Notable mentee feedback included the formation of an immediate connection with a peer supporter and feelings of "automatic trust" even after previously seeing a mental health professional for their care. Mentors described their participation in peer programs as a source for continued learning and inspiration for their own recovery.

One-to-one peer support is a cost-effective, well-received intervention that increases patient satisfaction and objective QOL measures across many fields. Outcome measurements of one-to-one peer mentorship programs have demonstrated high rates of patient satisfaction and positive psychological outcomes in patients suffering from diabetes, breast cancer, prostate cancer, colon cancer, and gynecologic cancers. The operating cost of peer support mentorship is low, and these programs can further relieve the health care system by reallocating access to patient support services to a community level.

ELIGIBILITY:
Inclusion Criteria:

* Eligible candidates will be English-speaking adults with non-metastatic facial skin cancers.

Exclusion Criteria:

* Candidates with severe symptoms of mood, anxiety, or substance use at time of recruitment screening. Participants who require interdisciplinary collaboration (e.g. MMS + plastic surgery, ENT, etc.) for treatment of their facial skin cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-10-12 (Actual); Primary Completion 2019-08-27 (Actual); Study Completion 2019-08-27 (Actual)

PRIMARY OUTCOMES:
Skin Cancer Index (SCI) scores | Enrollment
  Primary study measures include patient responses from the Skin Cancer Index (SCI), a disease-specific, 15-question validated QOL instrument. The SCI is divided into 3 subscales: appearance, emotion, and social domains. Higher scores indicate increased QOL.
Skin Cancer Index (SCI) scores | 1-week postoperative follow-up
  Primary study measures include patient responses from the Skin Cancer Index (SCI), a disease-specific, 15-question validated QOL instrument. The SCI is divided into 3 subscales: appearance, emotion, and social domains. Higher scores indicate increased QOL.
Skin Cancer Index (SCI) scores | 3-month postoperative follow-up
  Primary study measures include patient responses from the Skin Cancer Index (SCI), a disease-specific, 15-question validated QOL instrument. The SCI is divided into 3 subscales: appearance, emotion, and social domains. Higher scores indicate increased QOL.

SECONDARY OUTCOMES:
Qualitative participant feedback | 3-month postoperative follow-up
  Secondary measures will include a post study exit survey to evaluate participant satisfaction and program feedback via qualitative and quantitative variables.

CONTACTS AND LOCATIONS:
Locations (1):
- Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Guy GP Jr, Machlin SR, Ekwueme DU, Yabroff KR. Prevalence and costs of skin cancer treatment in the U.S., 2002-2006 and 2007-2011. Am J Prev Med. 2015 Feb;48(2):183-187. doi: 10.1016/j.amepre.2014.08.036. Epub 2014 Nov 10. PMID 25442229
- [Background] Zhang J, Miller CJ, O'Malley V, Etzkorn JR, Shin TM, Sobanko JF. Patient quality of life fluctuates before and after Mohs micrographic surgery: A longitudinal assessment of the patient experience. J Am Acad Dermatol. 2018 Jun;78(6):1060-1067. doi: 10.1016/j.jaad.2018.02.065. Epub 2018 Mar 5. PMID 29518455
- [Background] Sobanko JF, Zhang J, Margolis DJ, Etzkorn JR, Shin TM, Sarwer DB, Miller CJ. Patient-reported quality of life and psychosocial health prior to skin cancer treatment - A cross-sectional study. J Am Acad Dermatol. 2016 Jul;75(1):217-218.e2. doi: 10.1016/j.jaad.2016.01.033. No abstract available. PMID 27317520
- [Background] Sobanko JF, Sarwer DB, Zvargulis Z, Miller CJ. Importance of physical appearance in patients with skin cancer. Dermatol Surg. 2015 Feb;41(2):183-8. doi: 10.1097/DSS.0000000000000253. PMID 25654193
- [Background] Pearl RL, Shao K, Shin TM, Miller CJ, Sobanko JF. Acute Appearance Concerns in Patients Undergoing Mohs Surgery: A Single-Institution Cross-Sectional Study. Dermatol Surg. 2018 Oct;44(10):1349-1351. doi: 10.1097/DSS.0000000000001431. No abstract available. PMID 30256237
- [Background] Meyer A, Coroiu A, Korner A. One-to-one peer support in cancer care: a review of scholarship published between 2007 and 2014. Eur J Cancer Care (Engl). 2015 May;24(3):299-312. doi: 10.1111/ecc.12273. Epub 2014 Dec 16. PMID 25512107
- [Background] Badger K, Royse D. Adult burn survivors' views of peer support: a qualitative study. Soc Work Health Care. 2010;49(4):299-313. doi: 10.1080/00981380903493095. PMID 20379901